CLINICAL TRIAL: NCT06129461
Title: A Single Session Self-guided Acceptance-based Digital Intervention Targeting Food Cravings as Predictors of Disordered Eating in Pregnant People
Brief Title: A Single Session Self-guided Acceptance-based Digital Intervention Targeting Food Cravings in Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University at Albany (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Julia Hormes, Associate Professor, University at Albany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23E225
Record Dates: First submitted 2023-11-04; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Pregnancy Weight Gain; Eating Disorders; Perinatal Problems; Binge Eating; Craving
Keywords: gestational weight gain; loss of control eating; binge eating; food craving; mobile health intervention; single session intervention; Acceptance and Commitment Therapy
MeSH Terms: conditions — Gestational Weight Gain; Feeding and Eating Disorders; Bulimia | interventions — Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The intervention group will participate in a single-session, self-guided online intervention imparting skills grounded in Acceptance and Commitment Therapy. The one-hour workshop guides participants through evidence-based exercises, brief video clips, and reflection activities designed to clarify values and teach skills to foster acceptance, defusion, and present-moment awareness.
  Interventions: Behavioral: Single-session acceptance-based online workshop targeting food cravings as predictors of loss of control and binge eating in pregnancy
- Control (No Intervention): Participants in the control group will not receive any intervention; they will complete assessments on the same schedule as the intervention group (baseline, 1 month, at full term)

INTERVENTIONS:
Behavioral: Single-session acceptance-based online workshop targeting food cravings as predictors of loss of control and binge eating in pregnancy — Participants in the intervention will learn acceptance-based strategies for reducing the adverse impact of food cravings on eating behaviors. Unlike control-based strategies, acceptance-based strategies do not attempt to change the content or frequency of thoughts; rather, they foster willingness to acknowledge and experience uncontrollable thoughts, urges, and emotions as what they are - nothing more, nothing less. Acceptance-based approaches have demonstrated efficacy in reducing the adverse impact of food cravings on eating behaviors in non-pregnant samples.
  Arms: Treatment

SUMMARY:
Pregnancy is a time of heightened risk for disordered eating behaviors, which have been linked to adverse health outcomes in gestation, delivery, and the postpartum. These adverse outcomes may at least in part be mediated by greater risk of deviation from recommended gestational weight gain trajectories, especially in those engaged in binge and loss of control eating. This study will explore the efficacy of a single-session, self-guided online acceptance-based intervention targeting food cravings as powerful and modifiable predictors of binge and LOC eating in pregnancy.

DETAILED DESCRIPTION:
Pregnancy is a time of heightened risk for disordered eating behaviors, which have been linked to a range of adverse health outcomes in pregnancy, delivery, and the postpartum. These adverse outcomes may at least in part be mediated by greater rates of deviation from recommended weight gain trajectories, especially in those engaged in binge and loss of control eating. Food cravings are powerful triggers of binge and loss of control eating in non-pregnant populations with preliminary evidence linking cravings to disordered eating behaviors and greater weight gain in pregnancy as well. This study builds on preliminary evidence to suggest that acceptance-based approaches are effective in reducing the adverse impacts of cravings on behavior by exploring the efficacy of a single-session, self-guided online acceptance-based intervention targeting food cravings in pregnant participants as predictors of maladaptive eating behaviors and deviations from recommended gestational weight gain trajectories.

The efficacy of a single-session, self-guided online acceptance-based intervention targeting food cravings in pregnant participants will be examined in a randomized controlled trial. Pregnant individuals in the second trimester (n = 130) who endorse current cravings will be randomly assigned to the intervention or an untreated control group. The intervention group will participate in a single-session, self-guided online workshop imparting skills grounded in Acceptance and Commitment Therapy, including acceptance, defusion, and present-moment awareness. Both groups will complete comprehensive assessments at baseline, one-month follow-up, and at full-term. The results of this initial efficacy trial will inform the integration of acceptance-based self-guided health coaching targeting food cravings into routine prenatal care to prevent adverse outcomes associated with disordered eating behaviors in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Current residence in the United States
* Fluency in English
* Currently pregnant in the second trimester
* Experience of any food cravings

Exclusion Criteria:

* None beyond not meeting inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-11-14 (Estimated); Study Completion 2024-11-14 (Estimated)

PRIMARY OUTCOMES:
Prenatal Eating Behaviors Screening Tool | From study entry in 2nd trimester of pregnancy through delivery
  Eating disorder symptoms, including frequency of binge and loss-of-control eating
Gestational weight gain | From study entry in 2nd trimester of pregnancy through delivery
  Deviations from recommended gestational weight gain trajectories (in U.S. lbs)
Food Craving Questionnaire - Trait - Reduced | From study entry in 2nd trimester of pregnancy through delivery
  Frequency and intensity of food craving experiences

SECONDARY OUTCOMES:
Food Craving Acceptance and Action Questionnaire | Assessed at baseline and 1-month post-intervention
  Acceptance of and willingness to experience food cravings
Obsessive Compulsive Eating Scale | Assessed at baseline and 1-month post-intervention
  Intrusive thoughts and urges related to a craved target
White Bear Suppression Inventory | Assessed at baseline and 1-month post-intervention
  Thought suppression
Detail and Flexibility Questionnaire | Assessed at baseline and 1-month post-intervention
  Cognitive flexibility

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified and aggregate data may be made available to other researchers upon reasonable request.

REFERENCES:
- [Derived] Costello K, Timko CA, Anderson D, Hormes JM. Validation of the intolerance of uncertainty scale-12 in a sample of pregnant people. BMC Pregnancy Childbirth. 2025 Mar 27;25(1):363. doi: 10.1186/s12884-025-07434-1. PMID 40148844
- [Derived] Hormes JM, Timko CA. A clinical trial protocol of a single-session self-guided acceptance-based online intervention targeting food cravings as predictors of disordered eating in pregnant people. Contemp Clin Trials. 2024 May;140:107515. doi: 10.1016/j.cct.2024.107515. Epub 2024 Mar 26. PMID 38537903